CLINICAL TRIAL: NCT03432169
Title: Yoga vs Stretching in Veterans With Chronic Lower Back Pain: Does Mindfulness Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Dougherty, DC, Staff Chiropractor, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRBnet 1135250
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Yoga; Mindfulness

STUDY DESIGN:
Intervention Model Description: Group A receives Yoga (stretching with mindfulness) and Group B receives stretching (stretching without mindfulness)
Who Masked: Outcomes Assessor
Masking Description: Will code data entered into database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Active Comparator): Stretching with mindfulness
  Interventions: Other: Yoga (stretching plus mindfulness)
- Stretching (Active Comparator): Stretching exercises without mindfulness
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Yoga (stretching plus mindfulness) — Stretching plus mindfulness
  Arms: Yoga
Other: Stretching — Stretching alone
  Arms: Stretching

SUMMARY:
The purpose of this study is to demonstrate the feasibility of recruiting, enrolling and collecting outcome data on CLBP patients within the Veterans Affairs Community Based Rochester Outpatient Center who undergo an 8 week active exercise class with mindfulness (yoga) and without mindfulness (stretching class)

DETAILED DESCRIPTION:
The study will approach all new or existing patients within the chiropractic clinic between the ages of 18 and 89 who have low back pain greater than 12 weeks and pain greater than or equal to 3, who have no contraindications to active exercise. Patients will be queried as to interest and those interested will be consented. The investigators will recruit a total of 20 patients. Patients will then be randomized to receive either an 8 week active exercise class with mindfulness (yoga) or an 8 week active exercise class without mindfulness (stretching class). Both groups will have home exercise requirements and will be held accountable through the use of a home practice log. Outcomes will include: Pain (PEG), Quality of Life (PROMIS Global Health Survey GHS), Self Efficacy (2 Question), Fear Avoidance Belief, Castrophizing and Social Engagement. Outcomes will be collected at baseline, and again at the end of the 8 week intervention. Clinician open ended questionnaire will be given to both study clinicians at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veterans between the ages of 18-89
* Lower back pain > 12 weeks
* Have the ability to exercise independently.

Exclusion Criteria:

* Subjects will be excluded if
* They are currently enrolled in or maintain a home meditation practice
* If they are currently involved in a mindfulness or cognitive behavioral therapy group.
* If they have participated in a structured group yoga class in the last three months.
* If they have an open workers compensation or no-fault case or have undergone spinal surgery in the past 6 months.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  The main purpose of the study is to assess feasibility of conducting a larger trial. The study team will assess number of Veterans recruited and enrolled in the study. Number of sessions completed.

SECONDARY OUTCOMES:
PROMIS Global Health Scale (GHS): | baseline, immediately post intervention
  Patient reported outcome measurement information system has developed a quality of life tool that provides an overall index score for quality of life. This form has recently been validated in comparison to the EuroQual. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score always represents more of the concept being measured.
Pain, Engagement and General activity (PEG) | baseline, immediately post intervention
  An ultra-brief three-item scale derived from the Brief Pain Inventory (BPI), was a reliable and valid measure of pain among primary care patients with chronic musculoskeletal pain and diverse VA ambulatory patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester Outpatient Clinic (ROPC) of the Canandaigua VA Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No